CLINICAL TRIAL: NCT07086287
Title: Evaluation of the Efficacy of Recombinant Human Brain Natriuretic Peptide in Patients With Diuretic Resistance After Cardiac Surgery: a Prospective Single-center Single-blind Randomized Controlled Study
Brief Title: Evaluation of the Efficacy of rhBNP in Patients With Diuretic Resistance After Cardiac Surgery
Acronym: rhBNP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, GONG QIAN, Associate Chief Physician, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rhBNP with diuretic resistance
Record Dates: First submitted 2025-06-27; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: After Cardiac Surgery; Diuretic Resistance
Keywords: recombinant human brain natriuretic peptide; diuretic resistance; after cardiac surgery; the incidence of renal replacement therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhBNP group (Experimental): The rhBNP group was given positive inotropic agents, increased mean arterial pressure, restricted intake, and increased the dosage of diuretics. At the same time, rhBNP will be administered a venous loading dose of 1.5~2μg/kg, refer to the instructions for a maintenance dose of 0.0075-0.01μg/kg/min for continuous intravenous infusion for 72 hours.
  Interventions: Drug: rhBNP and standard basic treatment
- control group (No Intervention): The control group was given positive inotropic agents, increased mean arterial pressure, restricted intake, and increased the dosage of diuretics without rhBNP.

INTERVENTIONS:
Drug: rhBNP and standard basic treatment — After administering a bolus of rhBNP at 1.5-2 μg/kg intravenously, a maintenance dose of 0.0075-0.01 μg/kg/min is continuously infused intravenously for 72 hours, with the dosage adjusted based on blood pressure and heart rate; the control group receives standard basic treatment.
  Arms: rhBNP group

SUMMARY:
evaluation of the efficacy of recombinant human brain natriuretic peptide in patients with diuretic resistance after cardiac surgery: a prospective single-center single-blind randomized controlled study

DETAILED DESCRIPTION:
Postoperative adult patients (aged ≥18 years) with fluid overload were randomly assigned to groups, divided into the rhBNP group and the control group. The control group received positive inotropic agents, increased mean arterial pressure, restricted fluid intake, and increased the dosage of diuretics. The rhBNP group received conventional treatment in addition to a loading dose of 1.5-2 μg/kg intravenously, according to the instructions, to maintain a dosage of 0.0075-0.01 μg/kg/min continuously infused via intravenous pump for 72 hours, with dosage adjusted based on blood pressure. The grouping of subjects was concealed, and researchers were not allowed to access grouping information before the analysis was completed, with early unblinding prohibited. The primary research endpoint was the incidence of renal replacement therapy. Secondary research endpoints included the duration of tracheal intubation after cardiac surgery, CICU time after cardiac surgery, and length of hospitalization after cardiac surgery. Blood and urine samples were collected at the time of enrollment, 1 hour after maintaining the rhBNP dosage of 0.0075-0.01 μg/kg/min, and at 24 hours, 48 hours, and 72 hours after medication administration.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adult patients after cardiac surgery (age ≥ 18 years) (2) Fluid overload (3) Diuretic resistance Definition: Daily intravenous use of furosemide at a dose ≥ 80mg or equivalent doses of other diuretics, yet still unable to achieve an adequate urine output of 0.5~1.0mL/kg/h. Conversion formula for different loop diuretics: Oral furosemide 80mg = Intravenous furosemide 40mg = Oral/Intravenous torsemide 20mg = Oral/Intravenous bumetanide 1mg (4) Willing to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* (1) Preoperative CKD patients undergo regular dialysis treatment; (2) Postoperative use of CRRT; (3) Drug allergies involved in this study; (4) Those with corrected systolic blood pressure still < 90 mmHg after vasopressor use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of renal replacement therapy | From enrollment to discharge: at enrollment, the maintenance dose of rhBNP is 0.0075-0.01ug/kg/min, after 1 hour, 24 hours, 48 hours, and 72 hours post-medication.
  Indications for initiating renal replacement therapy (RRT): (1) Severe electrolyte disturbances, such as blood potassium >6.5 mmol/L with ECG abnormalities, or ineffective drug treatment; (2) Metabolic acidosis, pH <7.15 and HCO₃-<12 mmol/L, excluding respiratory factors; (3) Volume overload, pulmonary edema/persistent heart failure, and unresponsive to diuretics (e.g., urine output <200ml/2h during furosemide stress test positive); (4) Toxin removal, rhabdomyolysis (creatine kinase (CK) > 5000 U/L with acute kidney injury).

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
2030-01-01 Publication of academic papers
Supporting Information: Study Protocol
Time Frame: Starting from 2023-01-01, permanently.
Access Criteria: Access researchers from the China Clinical Trial Registry or clinicaltrials.gov .
URL: https://www.chictr.org.cn/

REFERENCES:
- [Result] Kourek C, Briasoulis A, Giamouzis G, Skoularigis J, Xanthopoulos A. Lyophilized recombinant human brain natriuretic peptide: A promising therapy in patients with chronic heart failure. World J Clin Cases. 2023 Dec 26;11(36):8603-8605. doi: 10.12998/wjcc.v11.i36.8603. PMID 38188212
- [Result] Li X, Wang R, Sun D, Yao Y, Wang T, Luo G, Liu M, Xu J, Cheng Z, Gao Q, Wang Y, Wu C, Xu G, Lv T, Zou J, Yan M. Risk Factors for Hypocoagulability After Cardiac Surgery: A Retrospective Study. Clin Appl Thromb Hemost. 2023 Jan-Dec;29:10760296231209927. doi: 10.1177/10760296231209927. PMID 37933155
- [Result] Thanavaro J, Taylor J, Vitt L, Guignon MS. Predictors and Outcomes of Acute Kidney Injury after Cardiac Surgery. Nephrol Nurs J. 2019 Jan-Feb;46(1):31-40. PMID 30835094
- [Result] Gong B, Wu Z, Li Z. Efficacy and safety of nesiritide in patients with decompensated heart failure: a meta-analysis of randomised trials. BMJ Open. 2016 Jan 6;6(1):e008545. doi: 10.1136/bmjopen-2015-008545. PMID 26739721
- [Result] Yancy CW, Krum H, Massie BM, Silver MA, Stevenson LW, Cheng M, Kim SS, Evans R; FUSION II Investigators. Safety and efficacy of outpatient nesiritide in patients with advanced heart failure: results of the Second Follow-Up Serial Infusions of Nesiritide (FUSION II) trial. Circ Heart Fail. 2008 May;1(1):9-16. doi: 10.1161/CIRCHEARTFAILURE.108.767483. PMID 19808265
- [Result] Wang H, Li Y, Chai K, Long Z, Yang Z, Du M, Wang S, Zhan S, Liu Y, Wan Y, Wang F, Yin P, Li W, Liao Y, Dong Y, Li X, Zhou J, Yiu KH, Zhou M, Huo Y, Yang J. Mortality in patients admitted to hospital with heart failure in China: a nationwide Cardiovascular Association Database-Heart Failure Centre Registry cohort study. Lancet Glob Health. 2024 Apr;12(4):e611-e622. doi: 10.1016/S2214-109X(23)00605-8. PMID 38485428
- See also: China Clinical Trial Registration Center — https://www.chictr.org.cn/
- Available data/document: Study Protocol: rhBNP — https://www.chictr.org.cn/ — China Clinical Trial Registration Center